CLINICAL TRIAL: NCT00609817
Title: An Open-Label Phase 1/2 Study of the Safety and Efficacy of GCS-100 in Subjects With Relapsed or Relapsed/Refractory Multiple Myeloma
Brief Title: Safety and Efficacy Study of GCS-100LE in the Treatment of Multiple Myeloma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Lack of funding
Sponsor: La Jolla Pharmaceutical Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PR-CS009
Record Dates: First submitted 2008-01-24; First posted 2008-02-07 (Estimated); Last update posted 2013-06-25 (Estimated); Status verified 2013-06

CONDITIONS: Multiple Myeloma
Keywords: Relapsed Multiple Myeloma; Refractory Multiple Myeloma; GCS 100
MeSH Terms: conditions — Multiple Myeloma | interventions — GCS-100; Bortezomib; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- GCS-100 (Experimental)
  Interventions: Drug: GCS-100; Drug: Bortezomib/Dexamethasone

INTERVENTIONS:
Drug: GCS-100 — GCS-100 160mg/m2 IV (in the vein) on Study Days 1, 4, 8 and 11 for up to 12 consecutive 21-day treatment cycles. Three patients will be assigned to each cohort until maximum tolerated dose is reached. The dose levels: 1) 160 mg/m2; 2) 210 mg/m2; 3) 280 mg/m2; 4) 370 mg/m2
Drug: Bortezomib/Dexamethasone — Bortezomid 1.3 mg/m2 and dexamethasone 20 mg/day plus an additional 20 mg of dexamethasone on the day following each of the GCS-100/bortezomib and dexamethasone dosing. GCS-100/bortezomib and dexamethasone dosed on Study Days 1, 4, 8 and 11 of each 21-day cycle after disease progression is noted.
  Other Names: Velcade; Decadron

SUMMARY:
A Phase 1, open-label, dose escalation, multi-center study in patients who have been diagnosed with multiple myeloma and who have relapsed or have refractory/relapsed disease after treatment with at least 2 prior therapies.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the safety and the dose-limiting toxicities of GCS-100 in subjects with relapsed or relapsed/refractory multiple myeloma, and to identify the maximum tolerated dose and/or the recommended dose for further studies.

The secondary objectives of this study are (i) to evaluate the safety of treatment with GCS-100 in combination with bortezomib (VelcadeTM) in subjects whose disease has progressed on GCS-100 alone; (ii) to evaluate the response to GCS-100 alone, in combination with bortezomib in subjects whose disease has progressed on GCS-100 alone, and during dexamethasone therapy in combination with GCS 100 plus bortezomib in subjects whose disease has progressed on GCS-100 plus bortezomib; (iii) to evaluate the utility of potential surrogate markers; (iv) to perform exploratory correlative analyses of bone marrow samples to define better the mechanisms of action and response to therapy.

ELIGIBILITY:
Inclusion Criteria:

* Subject is capable of understanding the purpose and risks of the study and is able to provide written Informed Consent.
* Subject is male or female, aged at least 18 years.
* Subject was diagnosed previously with multiple myeloma based on standard criteria.
* Subject has relapsed or relapsed/refractory disease following at least 2 prior therapies and/or lines of therapy (i.e., pre-planned comprehensive treatment regimens). Previously allogeneic and autologous bone marrow transplants, and prior therapy with bortezomib, are permitted.
* Subject's Karnofsky performance status is ≥ 60%.
* Subject's life expectancy is at least 3 months.
* Female subjects of childbearing potential (i.e., women who have not been surgically sterilized or have not been post-menopausal for at least 1 year), and male subjects with partners of childbearing potential, must agree to use medically acceptable methods of contraception throughout the study period.
* Subject is willing and able to comply with the prescribed treatment protocol and evaluations.

Exclusion Criteria:

* Subject is receiving concomitant medications (with the exception of bisphosphonates, erythropoietin, and/or up to 10 mg per day of prednisone, and with the exception of up to 100 mg hydrocortisone administered as premedication prior to administration of certain medications or blood products) and/or other therapy that may be active against multiple myeloma. Concurrent radiation therapy is not permitted.
* Subject received chemotherapy or other anti-cancer therapy that may be active against multiple myeloma within the 3 weeks prior to Study Day 1, and/or subject received nitrosureas within the 6 weeks prior to Study Day 1.
* Subject has not recovered from all toxic effects of previous chemotherapy, radiation therapy, biologic therapy, and/or experimental therapy.
* Subject received an investigational therapy within the 3 weeks prior to Study Day 1.
* Subject's clinical laboratory values met any of the following criteria within the 7 days prior to Study Day 1:

  1. Platelet count < 50,000 cells/mm3
  2. Absolute neutrophil count < 1,000 cells/mm3
  3. Hemoglobin < 8.0 g/dL (hemoglobin may be maintained by erythropoietin or transfusion)
  4. AST and/or ALT > 2.5 X the upper limit of normal
  5. Total bilirubin > 1.5 X the upper limit of normal
  6. Serum creatinine > 2 mg/dL
* Subject has a known history of human immunodeficiency virus (HIV), hepatitis B, and/or hepatitis C infection.
* Subject has a clinically relevant active infection and/or a serious co-morbid medical condition such as recent myocardial infarction, unstable angina, difficult-to-control congestive heart failure, uncontrolled hypertension, difficult-to-control cardiac arrhythmias, chronic obstructive or chronic restrictive pulmonary disease, and/or cirrhosis.
* Subject had major surgery within the 4 weeks prior to Study Day 1.
* Subject had another malignancy within the 3 years prior to study entry, with the exception of adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, in situ breast cancer, in situ prostate cancer, or other cancer for which the subject has been disease-free for at least the past 3 years.
* If female, subject is pregnant or breastfeeding.
* Subject has a known hypersensitivity to bortezomib, boron, and/or mannitol.
* Subject has a concomitant disease or condition, including laboratory abnormalities, which in the opinion of the Investigator could interfere with the conduct of the study or could put the subject at unacceptable risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2008-05; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
To evaluate GCS-100 related dose-limiting toxicity and to identify the maximum tolerated dose and/or the recommended dose for further studies. | Up to 12 consecutive 21-day treatment cycles

SECONDARY OUTCOMES:
To evaluate the safety of treatment with GCS-100 in combination with bortezomib (VelcadeTM) and dexamethasone in subjects whose disease has progressed on GCS-100 alone. | Up to 12 consecutive 21-day treatment cycles

CONTACTS AND LOCATIONS:
Overall Officials: Robert Schlossman, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (3):
- United States (3):
  - University of Florida, Gainesville, Florida
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Froedtert & Medical College Clinics, Medical College of Wisconsin, Milwaukee, Wisconsin